CLINICAL TRIAL: NCT00200551
Title: A Prospective, Randomized, Open, Multicentric Study Intended to Evaluate the Efficacy and Tolerability of Sequential Treatment Based on Rabbit Anti-T-lymphocyte Serum, of Mycophenolate Mofetil and of Cyclosporin, Without Concomitant Corticosteroids, After a First Cadaveric Renal Transplant
Brief Title: A Study of Mycophenolate Mofetil and Cyclosporin, Without Concomitant Corticosteroids, After a First Renal Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/00/6-G
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Renal Transplantation
MeSH Terms: interventions — Cyclosporine; Mycophenolic Acid; Antilymphocyte Serum; Adrenal Cortex Hormones

INTERVENTIONS:
Drug: Cyclosporin, mycophenolate mofetil, antilymphocyte serum and corticoids.
Drug: Cyclosporin, mycophenolate mofetil, antilymphocyte serum without corticoids.

SUMMARY:
The trial is planned as a multicentric, randomized, prospective, open study in accordance with a 1/1 plan, on parallel groups and 2 arms of treatment. A total of 200 patients with chronic renal insufficiency, included in the French national waiting list of the Establishment Français des Greffes [French Transplants Institution] and receiving a first renal transplant will be included, after signed agreement, in this study. All the patients will receive organs taken from brain-dead subjects. The patients will be given immunosuppressant treatment based on rabbit anti-T lymphocyte serum, CellCeptÒ and NeoralÒ cyclosporin. One group of 100 randomised patients will be given standard corticosteroid therapy as well during the first six months following the transplant. This group will be compared with a second group of 100 randomised patients who will be given a single dose of corticosteroids. The main aim of this study is to evaluate the number of acute rejection episodes in patients given a first renal transplant and subjected to an immunosuppressant protocol not containing corticosteroids. The hypothesis which is proposed is that, in the absence of corticosteroids and/or calcineurin inhibitors (i.e. cyclosporin and tacrolimus), antilymphocyte serum results in a certain state of "tolerance" in respect of the allograft. The second objective concerns the beneficial effect which the absence of corticosteroids may have on short- and long-term postoperative morbidity and mortality. One may in fact assume that the absence of corticosteroids will result in an extension of the transplant patient's life expectancy as a result of the reduction in cardiovascular complications. Cardiovascular complications are the most frequent cause of death after a renal transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is a candidate for a first cadaver renal transplantation and included on the national list of the Etablissement Français des Greffes
* Man or woman aged between 18 and 65 years
* Women of reproductive age must agree to use a reliable contraceptive method throughout the first year of the study
* Donor aged between 18 and 65 years
* Patient who has been given full information about the study and who has given his written informed consent to take part in it.

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Patient with an immunological risk considered high and defined as a percentage of anti-HLA antibodies of ³20% (previous or recent determination of T lymphocytes)
* Patient with a history of allergy to rabbit proteins
* Cold ischaemia time of more than 36 hours
* Patient allergic to macrolide antibiotics, to tacrolimus or to MMF
* Patient on immunosuppressant treatment before transplantation
* Patient suffering from a malignant neoplasm or with a history of malignant neoplasia, with the exception of treated baso- or spinocellular cancers
* Patient waiting for another transplant in addition to the kidney
* Patient who has already received an organ or tissue graft
* Leukocyte count <2000/mm3 and/or platelet count <50 000/mm3
* Patient suffering from focal glomerulonephritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2001-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the number of acute rejection episodes during the first year after transplantation in patients given a first renal transplant and subjected to an immunosuppressant protocol not containing corticosteroids.

SECONDARY OUTCOMES:
Clinical tolerance of the treatment with antilymphocyte
Any complication related to the corticosteroid treatment
Graft survival at 1, 2, 3, 4 and 5 years
Patient survival at 1, 2, 3, 4 and 5 years
Incidence of infectious and tumoral complications at 1, 2, 3, 4 and 5 years
Incidence of cardiovascular complications at 1, 2, 3, 4 and 5 years
Incidence of metabolic and lipid disorders at 1, 2, 3, 4 and 5 years
Bone osteodensitometry and folic acid levels before transplantation and at 2 weeks, 3 and 6 month after transplantation; then yearly up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Diego CANTAROVICH, MD, Principal Investigator — Nantes UH
Locations (5):
- France (5):
  - Besançon Universitary Hospital, France, Besançon
  - Montpellier Universitary Hospital, Montpellier
  - Nantes University Hospital, Nantes
  - Nice Universitary Hospital, Nice
  - Strasbourg Universitary Hospital, Strasbourg

REFERENCES:
- [Derived] Cantarovich D, Rostaing L, Kamar N, Saint-Hillier Y, Ducloux D, Mourad G, Garrigue V, Wolf P, Ellero B, Cassuto E, Albano L, Soulillou JP; FRANCIA Study Trial Investigators Group. Corticosteroid avoidance in adult kidney transplant recipients under rabbit anti-T-lymphocyte globulin, mycophenolate mofetil and delayed cyclosporine microemulsion introduction. Transpl Int. 2010 Mar 1;23(3):313-24. doi: 10.1111/j.1432-2277.2009.00971.x. Epub 2009 Oct 19. PMID 19843296